CLINICAL TRIAL: NCT04696653
Title: Using an Innovative Quality Improvement Process to Increase Delivery of Evidence-based Cardiovascular Risk Factor Care in Community Mental Health Organizations
Brief Title: A Quality Improvement Process to Support Delivery of Cardiovascular Care in Community Mental Health Organizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00269855; P50MH115842 (NIH)
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Hypertension; Dyslipidemias
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive unit based safety (CUSP) intervention arm (Other): CUSP is a quality improvement strategy developed by the Johns Hopkins University Armstrong Institute for Patient Safety and Quality that is used to improve care delivery.
  Interventions: Other: Comprehensive Unit Based Safety Program (CUSP)

INTERVENTIONS:
Other: Comprehensive Unit Based Safety Program (CUSP) — CUSP is a quality improvement strategy developed by the Johns Hopkins University Armstrong Institute for Patient Safety and Quality that is used to improve care delivery.

SUMMARY:
This pilot study will examine whether an implementation strategy will improve delivery of evidence-based care for cardiovascular risk factors for people with serious mental illness.

DETAILED DESCRIPTION:
In this pilot study, the investigators will work with health home programs and pilot test an adapted Comprehensive Unit Safety Program (CUSP) implementation strategy to improve mental health providers' delivery of evidence-based cardiovascular risk factor care for hypertension, dyslipidemia and diabetes for individuals with serious mental illness. The project will also characterize implementation processes, organizational and provider-level factors, and cardiovascular disease risk factor care and control.

ELIGIBILITY:
Inclusion Criteria:

Study population 1:

* Psychiatric rehabilitation program and health home team staff, including providers and leadership are those employed by the psychiatric rehabilitation program or health home program.
* English-speaking.

Study population 2:

* People with serious mental illness participating in psychiatric rehabilitation health home programs.
* English-speaking

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Daumit, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Adult Psychiatric Rehabilitation Program, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy KA, Gennusa J, Dalcin AT, Cook C, Goldsholl S, Fink T, Daumit GL, Wang NY, Thompson D, McGinty EE. Pilot of a team-based quality improvement strategy to improve cardiovascular risk factors care in community mental health centers. Front Psychiatry. 2025 Jan 31;16:1446985. doi: 10.3389/fpsyt.2025.1446985. eCollection 2025. PMID 39958153
- [Derived] McGinty EE, Thompson D, Murphy KA, Stuart EA, Wang NY, Dalcin A, Mace E, Gennusa JV 3rd, Daumit GL. Adapting the Comprehensive Unit Safety Program (CUSP) implementation strategy to increase delivery of evidence-based cardiovascular risk factor care in community mental health organizations: protocol for a pilot study. Implement Sci Commun. 2021 Mar 4;2(1):26. doi: 10.1186/s43058-021-00129-6. PMID 33663620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 85 participants (health home staff) were enrolled from 5 behavioral health home programs. The behavioral health home programs had a total of 498 health home clients (not enrolled) with data that was included in the analysis.
Units Other Than Participants: health home programs
Period: Overall Study
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Started | 85; 5 health home programs
Health Home Clients (Not Enrolled) | 498; 5 health home programs
Completed | 64; 5 health home programs
Not Completed | 21; 0 health home programs
Not completed — left organization | 18
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 16
  White | 61
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85
Comprehensive Unit Safety Program (CUSP) team membership [Count of Participants; unit: Participants] | 22

OUTCOME MEASURES:

1. Primary Outcome: Quality Improvement Culture as Assessed by the Modified Version of the Validated Survey on Patient Safety
Description: Each of the items in the modified survey is scored individually on 1-5 Likert scales. An average score is calculated by summing responses across all items and dividing by the total number of items. The average score ranges from 1-5. A higher average score signifies an organizational culture that is more supportive of quality improvement.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 3.8 (0.7)
  12 Month | 3.8 (0.6)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = 0, 95% CI 2-sided [-0.2 to 0.1]

2. Primary Outcome: Self-efficacy as Assessed by an Adapted Version of Compeau & Higgins' Task-focused Self-efficacy Scale
Description: Each of the items (Hypertension, Dyslipidemia, Diabetes) are scored individually on a 1-10 Likert scale, where 1=not at all confident and 10=totally confident. An average score is calculated by summing responses across all items and dividing by the total number of items. The average score ranges from 1-10. A higher score signifies greater self-efficacy.
Time Frame: Baseline, 12 Months
Population: CUSP team members with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 22
score on a scale
  Hypertension - Baseline | 6.0 (2.3)
  Hypertension - 12 Months | 7.1 (1.2)
  Dyslipidemia - Baseline | 5.9 (2.4)
  Dyslipidemia - 12 Months | 7.0 (1.4)
  Diabetes - Baseline | 6.2 (2.6)
  Diabetes - 12 Months | 7.3 (1.4)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; hypertension; Test type: Superiority; Mean Difference (Net) = 1.0, 95% CI 2-sided [0.2 to 1.8]
Statistical Analysis 2: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; dyslipidemia; Test type: Superiority; Mean Difference (Net) = 1.1, 95% CI 2-sided [0.0 to 2.1]
Statistical Analysis 3: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; diabetes; Test type: Superiority; Mean Difference (Net) = 1.0, 95% CI 2-sided [0.1 to 2.0]

3. Secondary Outcome: Acceptability as Assessed by the Acceptability of Intervention Measure
Description: Validated 4-item instrument measuring intervention acceptability of the Evidence based practice and CUSP strategy using the Acceptability of Intervention Measure. Each of the items will be measured on a 5-point Likert scale, where 1=completely disagree and 5=completely agree. An average score is calculated by summing responses across all items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater acceptability.
Time Frame: Baseline, 12 Months
Population: CUSP team members with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 19
score on a scale
  Evidenced Based Practice - Baseline | 4.4 (0.5)
  Evidenced Based Practice - 12 Months | 4.2 (0.5)
  CUSP Strategy - Baseline | 4.4 (0.5)
  CUSP Strategy - 12 Months | 4.2 (0.6)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Evidenced based practice; Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.1]
Statistical Analysis 2: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; CUSP strategy; Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.1]

4. Secondary Outcome: Appropriateness as Assessed by the Intervention Appropriateness Measure
Description: Four item instrument measuring intervention appropriateness of Evidence based practice and CUSP strategy using the Intervention Appropriateness Measure. Each of the items will be measured on a 5-point Likert scale, where 1=completely disagree and 5= completely agree. An average score is calculated by summing responses across all items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater appropriateness.
Time Frame: Baseline, 12 Months
Population: CUSP team members with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 19
score on a scale
  Evidenced Based Practice - Baseline | 4.3 (0.5)
  Evidenced Based Practice - 12 Months | 4.2 (0.7)
  CUSP Strategy - Baseline | 4.4 (0.5)
  CUSP Strategy - 12 Months | 4.2 (0.7)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; CUSP strategy; Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.2]
Statistical Analysis 2: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Evidenced based practice; Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

5. Secondary Outcome: Feasibility as Assessed by the Feasibility of Intervention Measure
Description: Four item instrument measuring intervention feasibility of Evidence based practice and CUSP strategy using the Feasibility of Intervention Measure. Each of the items will be measured on a 5-point Likert scale, where 1=completely disagree and 5=completely agree. An average score is calculated by summing responses across all items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater feasibility.
Time Frame: Baseline, 12 Months
Population: CUSP team members with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 19
score on a scale
  Evidenced Based Practice - Baseline | 4.3 (0.4)
  Evidenced Based Practice - 12 Months | 4.2 (0.6)
  CUSP Strategy - Baseline | 4.3 (0.4)
  CUSP Strategy - 12 Months | 4.2 (0.6)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; evidenced based practice; Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 2: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; CUSP strategy; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.2]

6. Secondary Outcome: Clients With Hypertension Control
Description: Measured with blood pressure (BP) readings reported by staff . Clients with control defined as a BP <130/80 mmHg.
Time Frame: Baseline and 12 Months
Population: Clients identified as having hypertension with collected blood pressure reading at either baseline or 12 months were analyzed under modeling approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 224
Participants
  Baseline | 41
  12 Months | 59
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.9 to 2.2]

7. Secondary Outcome: Clients With Dyslipidemia Control
Description: Measured with cholesterol readings reported by staff. Clients with controlled dyslipidemia defined as total cholesterol <200 mg/dL and low-density lipoprotein (LDL) <130 mg/dL.
Time Frame: Baseline and 12 Months
Population: Clients identified as having dyslipidemia with collected lipid data at either baseline or 12 months were analyzed under modeling approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 158
Participants
  Baseline | 70
  12 Months | 75
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.1 to 1.9]

8. Secondary Outcome: Clients With Diabetes Control
Description: Measured using HbA1c tests reported by staff . Clients with controlled diabetes defined as HbA1c<7.0.
Time Frame: Baseline and 12 Months
Population: Clients identified as having diabetes with collected HBA1c at either baseline or 12 months were analyzed under modeling approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 119
Participants
  Baseline | 53
  12 Months | 55
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.4]

9. Secondary Outcome: Clients Diagnosed With Diabetes Mellitus Who Received HBA1c Measurement
Description: The number of clients who have a HBA1c measurement reported by the participating staff.
Time Frame: Baseline and 12 Months
Population: Clients identified as having diabetes at either baseline or 12 months were analyzed under modeling approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 145
Participants
  Baseline | 92
  12 Months | 99
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.2 to 2.6]

10. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Diabetes Mellitus Who Received a Lipid Panel
Time Frame: Baseline, 6 and 12 months
Population: This data was supposed to be sourced from the electronic health record of participating sites. Sites did not collect this data, and the study is now completed so there will be no future data collection
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Diabetes Mellitus Who Received Statin Therapy
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 10
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Diabetes Mellitus Who Received a Dilated Eye Exam
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 10
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Diabetes Mellitus Who Received a Foot Exam
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 10
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

14. Secondary Outcome: Clients Diagnosed With Dyslipidemia Who Received a Lipid Panel
Description: The number of clients who have a lipid panel reported by the participating staff.
Time Frame: Baseline and 12 Months
Population: Clients identified as having dyslipidemia at either baseline or 12 months were analyzed under modeling approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 213
Participants
  Baseline | 131
  12 Months | 133
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Odds Ratio (OR) = 1.2, 95% CI 2-sided [1.0 to 1.6]

15. Secondary Outcome: Teamwork Within Teams as Assessed by the Implementation Climate Scale
Description: Four items measuring teamwork. Each of the items will be measured on a 5-point Likert scale, where 1=strongly disagree and 5=strongly agree. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies better teamwork within units.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 4.1 (0.9)
  12 Months | 4.0 (0.8)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]

16. Secondary Outcome: Supervisor/Manager Expectations and Actions Promoting Quality as Assessed by the Implementation Climate Scale
Description: Four items measuring the degree to which a provider's supervisor promotes quality improvement. Each of the items will be measured on a 5-point Likert scale, where 1=strongly disagree and 5=strongly agree. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater promotion of quality improvement.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 4.0 (0.9)
  12 Months | 4.1 (0.8)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

17. Secondary Outcome: Organizational Learning Assessed by the Implementation Climate Scale
Description: Three items measuring organizational learning environment. Each of the items will be measured on a 5-point Likert scale, where 1=strongly disagree and 5=strongly agree. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater organizational learning.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 3.9 (0.8)
  12 Months | 3.9 (0.6)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.1]

18. Secondary Outcome: Management Support for Patient Safety as Assessed by the Implementation Climate Scale
Description: Three items measuring the degree to which organization management supports quality improvement. Each of the items will be measured on a 5-point Likert scale, where 1=strongly disagree and 5=strongly agree. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater management support for quality improvement.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 3.7 (1.0)
  12 Months | 3.7 (0.8)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

19. Secondary Outcome: Overall Perceptions of Quality Improvement Culture as Assessed by the Implementation Climate Scale
Description: Three items measuring the perception's of the organization's quality improvement culture. Each of the items will be measured on a 5-point Likert scale, where 1=strongly disagree and 5=strongly agree. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies better quality improvement culture.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 3.7 (0.9)
  12 Months | 3.6 (0.8)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.0]

20. Secondary Outcome: Feedback and Communication About Error as Assessed by the Implementation Climate Scale
Description: Three items measuring feedback and communication about quality improvement. Each of the items will be measured on a 5-point Likert scale, where 1=never and 5=always. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies better feedback and communication.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 3.8 (0.9)
  12 Months | 3.7 (0.8)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.3 to 0.0]

21. Secondary Outcome: Communication Openness as Assessed by the Implementation Climate Scale
Description: Three items measuring perceptions of communication openness in the organization. Each of the items will be measured on a 5-point Likert scale, where 1=never and 5=always. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies better communication openness.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 3.5 (0.8)
  12 Months | 3.5 (0.8)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.3]

22. Secondary Outcome: Frequency of Events Reported as Assessed by the Implementation Climate Scale
Description: Three items assessing the degree to which mistakes are reported at the organization. Each of the items will be measured on a 5-point Likert scale, where 1=never and 5=always. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies more frequent mistake reporting.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 4.0 (0.9)
  12 Months | 4.1 (0.8)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.2]

23. Secondary Outcome: Teamwork Across Teams as Assessed by the Implementation Climate Scale
Description: Four items assessing teamwork across units. Each of the items will be measured on a 5-point Likert scale, where 1=strongly disagree and 5=strongly agree. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies better teamwork across units.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 3.9 (0.9)
  12 Months | 3.9 (0.8)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

24. Secondary Outcome: Staffing as Assessed by the Implementation Climate Scale
Description: Two items assessing staffing capacity. Each of the items will be measured on a 5-point Likert scale, where 1=strongly disagree and 5=strongly agree. An average score is calculated by summing responses across items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies better staffing capacity.
Time Frame: Baseline, 12 Months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 84
score on a scale
  Baseline | 2.9 (0.9)
  12 Months | 2.8 (0.9)
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.0]

25. Secondary Outcome: Clients With Hypertension Who Had a Blood Pressure Measurement
Description: The number of clients who have a blood pressure measurement reported by the participating staff.
Time Frame: Baseline and 12 Months
Population: Clients identified as having hypertension at either baseline or 12 months were analyzed under modeling approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 242
Participants
  Baseline | 166
  12 Months | 186
Statistical Analysis 1: Comparison: Comprehensive Unit Based Safety (CUSP) Intervention Arm; Test type: Superiority; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.0 to 3.3]

26. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Diabetes Mellitus Who Received a Urine-protein-creatinine Test
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 10
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

27. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Dyslipidemia Who Are on a Statin Medication
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 10
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

28. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Hypertension Who Received Lifestyle Counseling
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 10
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

29. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Diabetes Mellitus Who Received Lifestyle Counseling
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 10
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

30. Secondary Outcome: Change in the Percent of Individuals Diagnosed With Dyslipidemia Who Received Lifestyle Counseling
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 10
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse Events Not Collected
Arm/Group | Comprehensive Unit Based Safety (CUSP) Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT04696653/Prot_SAP_000.pdf